CLINICAL TRIAL: NCT02092415
Title: Assessment of Limb Perfusion During Junctional Tourniquet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Junctional Tourniquet
Record Dates: First submitted 2014-01-06; First posted 2014-03-20 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Bleeding
Keywords: Tourniquet; Muscle perfusion; Contrast ultrasound
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Normal subjects (Experimental): Normal subjects, all of whom undergo brief application of junctional tourniquet
  Interventions: Device: Application of a Junctional Tourniquet

INTERVENTIONS:
Device: Application of a Junctional Tourniquet — All subjects will be studied at baseline and after placement of a junctional tourniquet to the femoral artery.

SUMMARY:
The goal of this study is to use contrast enhanced ultrasound to determine the degree to which flow is reduced during application of a junctional tourniquet (JT). Contrast enhanced ultrasound is performed to quantify thigh and calf perfusion at baseline and during application of the JT

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Age 19-50

Exclusion Criteria:

* Peripheral artery disease
* Known heart failure
* Right to left shunt
* Pregnancy
* Presence of femoral artery aneurysm

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Lindner, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

REFERENCES:
- [Derived] Davidson BP, Belcik JT, Mott BH, Landry G, Lindner JR. Quantification of residual limb skeletal muscle perfusion with contrast-enhanced ultrasound during application of a focal junctional tourniquet. J Vasc Surg. 2016 Jan;63(1):148-53. doi: 10.1016/j.jvs.2014.06.107. Epub 2014 Jul 24. PMID 25065582

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Subjects
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Normal Subjects
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Muscle Perfusion
Description: Contrast ultrasound perfusion imaging will be performed at baseline and 1 min after application of the JT.
Time Frame: baseline and 1 min post occlusion
Measure: Mean (Standard Error); unit: IU/s
Groups:
- Normal Subjects Baseline Flow: Normal subjects, all of whom undergo brief application of junctional tourniquet
  Application of a Junctional Tourniquet: All subjects will be studied at baseline and after placement of a junctional tourniquet to the femoral artery.
- Normal Subjects - Tourniquet Flow: Perfusion measured at time of tourniquet placement
Arm/Group | Normal Subjects Baseline Flow | Normal Subjects - Tourniquet Flow
Number analyzed (Participants) | 10 | 10
IU/s | 0.32 (0.10) | 0.10 (0.03)

ADVERSE EVENTS:
Arm/Group | Normal Subjects
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No